CLINICAL TRIAL: NCT04332705
Title: Role of the Protozoa Cryptosporidium in the Development of Colorectal Cancer in Humans
Brief Title: Cryptosporidium Infection and Human Colorectal Cancer
Acronym: Crypto-K
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lille Catholic University (Other)
Collaborators: Institut Pasteur de Lille (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0091
Record Dates: First submitted 2020-03-31; First posted 2020-04-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Colonic Neoplasms; Cryptosporidiosis
Keywords: Colon cancer; Cryptosporidiosis; Prevalence; Infection and cancer
MeSH Terms: conditions — Colonic Neoplasms; Cryptosporidiosis; Infections; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Surgical specimens or biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with colon cancer: Patients with colon cancer of recent diagnosis will be recruited in consultation either in the surgical or gastroenterology departments
  Interventions: Diagnostic Test: Detection of Cryptosporidium infection
- Patients without colon cancer: Patients without colon cancer but with other gastrointestinal pathology needing a biopsy or a surgical procedure will be recruited either in the surgical or gastroenterology departments
  Interventions: Diagnostic Test: Detection of Cryptosporidium infection

INTERVENTIONS:
Diagnostic Test: Detection of Cryptosporidium infection — A biopsy or a surgical sample will be collected from every participant

SUMMARY:
It has been reported that Cryptosporidium parvum, a species of a protozoan frequently isolated from humans and animals, is able to induce digestive adenocarcinoma in a rodent model. Consistently, some epidemiological studies have reported an association with cryptosporidiosis in patients with colorectal adenocarcinoma. However, the correlation between cryptosporidiosis and human digestive cancer remains unclear at this time, and it is not known whether this intracellular parasite, considered an opportunistic agent, is able to induce gastrointestinal malignancies in humans. In order to add new arguments for a probable association between cryptosporidiosis and digestive human cancer, the main aim of this study is to determine prevalence and to identify species of Cryptosporidium among a French digestive cancer population.

ELIGIBILITY:
Inclusion Criteria:

Cases:

* Age ≥ 18 years old
* Patients with colonic adenocarcinoma/intraepithelial neoplasia diagnosed prior to chemotherapy or radiotherapy who will undergo scheduled surgery. Patients with rectal cancer with indication for neoadjuvant treatment will still be included, but only biopsies used for diagnosis will be used
* Patient capable of receiving informed information
* Written informed consent
* Affiliation to a social security scheme

Controls:

* Age ≥ 18 years old
* Patients with endoscopic indication for benign pathology
* Patients with indication for colectomy for benign pathology
* Patients with digestive cancer (stomach, oesophagus, biliary, pancreatic, etc.) of any type other than colorectal cancer before chemotherapy or radiotherapy
* Patient capable of receiving informed information
* Written informed consent
* Affiliation to a social security scheme

Exclusion Criteria:

* Patients undergoing pre-operative chemotherapy.
* Patients who have already had chemotherapy for less than one year or other immunosuppressive treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The cases will be the patients with colon cancer of recent diagnosis recruited in consultation either in the surgical or gastroenterology departments. The controls will be the patients without colon cancer but with other gastrointestinal pathology needing a biopsy or a surgical procedure and recruited either in the surgical or gastroenterology departments
Sampling Method: Non-Probability Sample
Enrollment: 324 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Cryptosporidium | 3 years
  A biopsy or a surgical sample will be collected from every participant which will be then screened for Cryptosporidium using a Polymerase chain reaction (PCR) in order to obtain a prevalence of positive individuals

SECONDARY OUTCOMES:
Rate of occurrence of parasite development in the tumoral zone (yes/no) compared to the peri-tumoral zone. | 3 years
  A biopsy or a surgical sample containing the tumoral and peri-tumoral areas will be collected only from the cases which will be then screened for Cryptosporidium using PCR
Significance of the association between the histological grade of the lesion and the Cryptosporidium species | 3 years
  Significance of the association between the histological grade defined by the Vienna classification of tumors and the species of Cryptosporidium and the Cryptosporidium species.The main species of Cryptosporidium infecting humans are C. parvum and C. hominis, however, other species can also infect humans.
Significance of the association between the histological grade of the lesion and the parasitic charge in tissues | 3 years
  Significance of the association between the histological grade defined by the Vienna classification of tumors and the species of Cryptosporidium and the parasitic charge in the tissues that will be determined by quantitative polymerase chain reaction (qPCR)
The rate of change in the expression or localization of certain markers known or suspected to be involved in the process of carcinogenesis. | 3years
  Some markers known to be associated to cancer development will be explored such as: Beta-catenin, P53, APC (adenomatous polyposis coli), etc.
The association between the rate of lymphocytes (CD3, CD4, CD8, CD19 and CD4/CD8 ratio) and the presence of parasites in biopsies or surgical specimens | 3 years
  Because Cryptosporidium is an opportunistic agent that causes significant morbidity and mortality in immunocompromised patients, it is possible that individuals with malignancies, have a higher risk of developing infection with this parasite, especially when their immunosuppression is more severe. To rule out this possibility this association will be determined.
Rate of development of a neoplastic lesion in the human explants | 3 years
  A three-dimensional culture model will be developed using colon samples from healthy tissues of several control patients. An experimental Cryptosporidium infection will be tested in order to determine the development of neoplastic lesions in these human explants.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Nunes, MD, Study Director — GHICL; Gabriela Certad, MD, PhD, Principal Investigator — GHICL
Locations (1):
- Groupement des Hôpitaux de l'Institut Catholique de Lille, Lomme, Nord, France